CLINICAL TRIAL: NCT04602455
Title: The Impact of Heartfulness Program on Loneliness in High School Students in the US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heartfulness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020/05/8
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Loneliness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heartfulness Group (Experimental): Participants were asked to practice relaxation tools for 15 minutes a day using the calendar and HeartBot app, and participate in once a week webinar for 30 minutes during the four weeks. UCLA Loneliness scale was recorded prior to the start of the study and at its end after the duration of 4 weeks. The score was reviewed to see the changes in the loneliness scale.
  Interventions: Behavioral: Self-Care Program through Heartfulness
- Control Group (No Intervention): The control group had no change in their daily routines.

INTERVENTIONS:
Behavioral: Self-Care Program through Heartfulness — A four-week Self-Care program through Heartfulness will be offered to participants in the Heartfulness group. This would include a daily practice of relaxation tools for 15 minutes a day using an app and once a week webinar for 30 minutes. Guided relaxation and meditation sessions will be offered to the participants during the intervention weeks. These virtual sessions were conducted by Heartfulness Champions and certified trainers from Heartfulness Institute.
  Arms: Heartfulness Group

SUMMARY:
This quantitative study assesses the baseline loneliness scores in all the high school students in the US. Assessments at baseline will include the UCLA loneliness scale. The Google form questionnaire will ask the high schoolers for their email address and their parent's email address (if they are under 18). The form will also include a question eliciting interest in participation in the 4-weeks Heartfulness program. The program will include tools that promote a heart-based nurturing environment focusing on relaxation, positivity, and developing growth mindsets.

DETAILED DESCRIPTION:
The specific aims of the study are:

1. To assess the current level of loneliness in high school students through the UCLA loneliness scale.
2. To assess the beneficial impact of the Heartfulness program on loneliness in high school students in the US.

ELIGIBILITY:
Inclusion Criteria:

* Participants are High School students in the US and willing to participate in the study

Exclusion Criteria:

* Non-English speaking high school students in the US and those with mental health diagnoses such as Major Depressive Disorder and Anxiety disorders.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Assess the current level of Loneliness | Baseline data through the pre-UCLA survey scores
  To assess the current level of loneliness in high school students through UCLA loneliness scale.
Changes in Loneliness levels | 28 days for 15 minutes every day based on a 28-day calendar
  To assess the beneficial impact of Heartfulness program on loneliness in high school students in the US.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjani B Iyer, PhD, Principal Investigator — Heartfulness Institute
Locations (1):
- Ranjani B Iyer, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publish a research paper with details on the study design, protocol, analysis of data, and report on implications to stress management and wellness tools.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting six months after publication
Access Criteria: Access criteria IPD and any additional supporting information will be shared with the researchers furthering research in stress management and emotional wellness tools.